CLINICAL TRIAL: NCT07212010
Title: Integrative Neurodevelopmental Approach to Cerebral Vision Impairment (CVI): Screening and Subtyping in Early Childhood
Brief Title: Neurodevelopmental Outcomes in Cerebral Visual Impairment
Acronym: CVI-ND
Status: Enrolling by invitation | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2024-0772; R01EY036154-01A1 (NIH)
Record Dates: First submitted 2025-09-22; First posted 2025-10-08 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Cerebral Visual Impairment
Keywords: Cerebral visual impairment; screening; Neurodevelopment; vision; cortical visual impairment
MeSH Terms: conditions — Blindness, Cortical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Screening: This group will be screened for CVI in the first year of life. Children with positive screens for CVI will undergo a comprehensive CVI evaluation.
- Neurodevelopment: Children in this group will participate in a multi-disciplinary CVI clinic as well as neurodevelopmental testing and a neuro-ophthalmic eye exam at baseline and 12 months later.

SUMMARY:
Cerebral visual impairment (CVI) is one of the leading causes of pediatric visual impairment and negatively impacts the development of motor, language, and cognitive skills. This study proposes to (1) establish a novel and easy to use CVI screening algorithm for infants and (2) develop CVI subtypes based on vision, motor, language, and cognition. The overarching goal is to identify CVI early and enhance our comprehension of CVI's impact on a child's development. The results will fundamentally change the approach to designing treatments for children with CVI.

DETAILED DESCRIPTION:
Cerebral visual impairment (CVI) is the leading cause of visual impairment in children. Although the onset is typically early in life, diagnosis is often delayed until preschool age or later. Early identification is critical for optimal development. Vision is essential in incidental and intentional learning used to build foundational motor, language, and cognitive skills. The proposed research aims to (1) develop a screening algorithm for early detection of CVI and (2) establish neurodevelopmental profiles that will inform intervention for children diagnosed with CVI. The overarching hypothesis is that early detection of CVI and understanding the relationship between visual impairment and neurodevelopment are imperative for creating interventions to optimize a child's abilities. In the first aim, a novel screening algorithm for CVI detection in infants will be tested at three time points between 4-12 months corrected age. In the second aim, an interdisciplinary standardized assessment protocol will be utilized, including visual and developmental evaluations at two time points to create neurodevelopmental subtypes in young children with CVI. This proposal will be implemented by an interdisciplinary research team with a well-established track record of clinical practice and research in CVI. This innovative proposal will lead to a paradigm shift in the current approach to CVI management in young children. The findings from this study will lead to the development of a screening protocol for early detection of CVI that can be easily incorporated into medical practice by providers who routinely interact with young infants and, in time, become standard practice. Additionally, the established neurodevelopmental profiles will serve as the cornerstone for creating comprehensive clinical protocols guiding the care and treatment of children diagnosed with CVI.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1 (CVI Risk Group): Infants 8 months of age and who meet any of the following:

  * The presence of any of the following comorbid diagnoses (CVI risk criteria): brain injury, hypoxia/ischemia, congenital structural abnormalities of the brain, genetic syndromes, epilepsy, infantile spasms/seizures, central nervous system infection, intrauterine drug/alcohol exposure, brain volume loss, or periventricular leukomalacia.
  * Presence of any of the following abnormal neuro-imaging findings (CVI risk criteria): Vascular insults, underlying genetic/structural/migrational abnormality, brain atrophy, prematurity sequelae, hydrocephalus, presumed metabolic findings, presumed infection findings.

Aim 1: (control group): Infants less than 8 months of age negative for CVI risk criteria (see above).

Exclusion Criteria: Aim 1: (both groups): Known visually impairing conditions of the eyes and optic nerves (e.g., inherited retinal diseases, bilateral moderate-to-severe optic nerve hypoplasia), cataracts, retinopathy of prematurity with significant visual sequelae (e.g. macular ectopia or retinal detachment) will be excluded from the study to ensure CVI is the primary cause of a positive PreViAs screen.

Aim 2: Inclusion criteria:

* Children 12-< 60 months of age
* Confirmed diagnosis of CVI

Children must meet at least 1 of these 2 criteria to confirm the diagnosis of CVI during a CVI clinic visit: I: (1) the presence of visual function impairment (e.g., visual acuity) not attributed to anterior visual pathway abnormalities (except mild optic atrophy) or 2) evidence of visual perception/functional vision deficit.

Aim 2: Exclusion Criteria:

* Children with autism spectrum disorder
* Children with ocular conditions including inherited retinal diseases, congenital cataracts, anterior segment dysgenesis, optic nerve hypoplasia, and retinopathy of prematurity with profound visual impairment due to anatomical abnormalities
* A chart review will take place to review for exclusion criteria. Children who are identified with one of these potential exclusion criteria will be formally evaluated/screened through a neuro-ophthalmology exam to confirm the presence or absence of the exclusionary diagnoses in the chart. This will occur prior to consenting and/or scheduling any other testing.

Ages: 6 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Aim 1: (at risk group) Children with medical and neuroimaging conditions that put children at high risk for cerebral visual impairment (control group) age matched peers without high-risk medical and neuroimaging conditions.
  Aim 2: Children with a diagnosis of cerebral visual impairment confirmed by a CVI multidisciplinary team visit.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Preverbal Visual Assessment (PreViAs) | Aim 1: 6, 9, and 12 months of age (corrected age if born preterm)
  The PreViAs (Preverbal Visual Assessment) is a questionnaire designed to assess visual cognitive behavior in infants under 24 months of age, through caregiver report. It consists of 30 questions that evaluate visual attention, communication, motor coordination, and processing skills. The questionnaire aims to identify visual difficulties that may not be detected through standard vision tests, allowing for early intervention and support for children at risk for visual impairments.
Visual Acuity | Aim 1: If/when visual concern are indicated on the Preverbal Visual Assessment (PreViAs) screening tool and/or at 12 months age (corrected if preterm); Aim 2: At enrollment (baseline) and 12 months later
  This study will offer several age and cognitively appropriate assessments to test visual acuity. Each child will participate in a visual acuity test. Optotype (recognition acuity) test of binocular visual acuity (Lea Number, Lea Symbol, or other Snellen equivalent) chart will be measured at a distance and near. Teller Acuity cards (grading resolution acuity) will be used with infants and young children who are nonverbal or pre-verbal and do not require a verbal response.
Contrast sensitivity | Aim 1: If/when visual concern are indicated on the Preverbal Visual Assessment (PreViAs) screening tool and/or at 12 months age (corrected if preterm); Aim 2: At enrollment (baseline) and 12 months later.
  This study will offer several assessments to test visual function depending on age and cognitive ability. Contrast sensitivity threshold is a measure of visual function. Contrast sensitivity will be measured by the Heiding Heidi cards using 2 alternative forced choice, Lea symbols or numbers flip chart, Peli Robson near chart.
Visual Fields | Aim 1: If/when visual concern are indicated on the Preverbal Visual Assessment (PreViAs) screening tool and/or at 12 months age (corrected if preterm); Aim 2: At enrollment (baseline) and 12 months later
  This study will offer several assessments to test the peripheral visual field depending on age and cognitive level. Assessing visual fields is a measure of visual function. Kinetic arc perimetry or confrontation visual field testing.
Color Vision | Aim 2: At enrollment (baseline) and 12 months later
  This study will offer several assessments to test color vision depending on age and cognitive level. The American Optical Hardy-Rand-Ritler (AO HRR) color plates using symbol detection or Panel 16 Quantitative Color Vision Test - Double Set (D-16) using chip alignment or matching paradigm.
Eye Motility | Aim 1: If/when visual concern are indicated on the Preverbal Visual Assessment (PreViAs) screening tool and/or at 12 months age (corrected if preterm); Aim 2: At enrollment (baseline) and 12 months later
  This study will offer several tests of eye motility depending on age and cognitive level. The following eye movements will be assessed by direct observation using developmentally appropriate targets: Fixation (absent, sporadic, unstable, stable); Smooth pursuit (absent, discontinuous, normal); Saccades (absent, hypometric, normal), and alignment to both distant and near targets. We will also measure eye gaze using a video-based eye tracking system.
Objects in motion | Aim 1: If/when visual concern are indicated on the Preverbal Visual Assessment (PreViAs) screening tool and/or at 12 months age (corrected if preterm); Aim 2: At enrollment (baseline) and 12 months later
  The ability to recognize objects that are in motion or the inability to recognize and/or attend to objects without motion. This will be assessed through clinical observation and parent report.
Accomodation | Aim 1: If/when visual concerns are indicated on the Preverbal Visual Assessment (PreViAs) screening tool and/or at 12 months of age (corrected if preterm); Aim 2: At enrollment (baseline) and 12 months later.
  Accommodative response will be measured through dynamic retinoscopy or the monocular estimation method.
Stereo Acuity | Aim 2: At enrollment (baseline) and 12 months later
  Stereoacuity will be administered at near (40cm) in current spectacle correction using the Randot Butterfly and Randot Preschool stereoacuity tests. Stereoacuity is defined as the smallest disparity in which the subject can correctly name or match at least 3 out of 4 target objects in the Randot Preschool stereoacuity tests.
Hemispatial neglect | Aim 2: At enrollment (baseline) and 12 months later
  Hemispatial neglect is measured when indicated using line bisection, Teddy Bear, and/or bell test.
Object recognition | Aim 2: At enrollment (baseline) and 12 months later.
  Formal and informal measures of object recognition are used. Formal measures include Lea Symbols (color puzzle, black and white puzzle, 2D representation). Informal measures include recognition of 2D and 3D materials, both near and at a distance.
Optic Ataxia | Aim 2: At enrollment (baseline) and 12 months later
  The LEA Mailbox test will be used to evaluate optic ataxia. The movements of the wrist and fingers are observed as the subject attempts to pass a card through the slot of a large, round disc. The ability of the subject to move the card towards the slot and to orient in the direction of the slot will be recorded. Alternatively, for younger participants, toys such as a piggy bank will be used.
Apraxia of the upper and lower limb | Aim 1: If/when visual concern are indicated on the Preverbal Visual Assessment (PreViAs) screening tool and/or at 12 months age (corrected if preterm); Aim 2: At enrollment (baseline) and 12 months later
  Upper limb apraxia is measured through clinical observation of hand and arm movement toward an object of interest. This measurement will begin at 4 months of age. Lower limb apraxia will be measured through clinical observation of foot and leg movement toward an object of interest. This will be measured starting at 12 months of age.
Spatial Perception | Aim 2: At enrollment (baseline) and 12 months later
  The ability to identify and match rectangles of different orientations and sizes using the Lea Rectangle game, shape sorter, or puzzles.
Simultanagnosia | Aim 2: At enrollment (baseline) and 12 months later
  The ability to attend to more than one object simultaneously will be assessed through clinical observation, AO HRR color plates, and birthday party test.
Facial Recognition | Aim 1: If/when visual concern are indicated on the Preverbal Visual Assessment (PreViAs) screening tool and/or at 12 months age (corrected if preterm); Aim 2: At enrollment (baseline) and 12 months later
  The ability to recognize familiar and/or unfamiliar faces will be assessed through parent report, 9-gaze app and NEPSY.
Facial Expressions | Aim 1: If/when visual concern are indicated on the Preverbal Visual Assessment (PreViAs) screening tool and/or at 12 months age (corrected if preterm); Aim 2: At enrollment (baseline) and 12 months later
  The ability to interpret facial expresssions will be measured through parent report and Lea expressions test (two-alternative forced choice)
Children's Visual Impairment Test (CVIT) | Aim 2: At enrollment (baseline) and 12 months later
  This study will offer several assessments to test functional vision depending on age and ability level. The Children's Visual Impairment Test (CVIT) 3-6 is a measure of visual function. The CVIT is a standardized, non-verbal assessment designed to evaluate visual perceptual abilities in children aged 3 to 6 years who may have visual impairments or developmental delays. It is an assessment of how well a child can recognize and match visual patterns, independent of language or motor skills. It is completed on the computer. The domains assessed include form perception, spatial relationships, and object recognition.
Beery-Buktenica Developmental test of Visual Motor Integration (Beery VMI) | Aim 2: At enrollment (baseline) and 12 months later
  This study will offer several assessments to test functional vision depending on age and ability level. The Beery-Buktenica Developmental Test of Visual-Motor Integration (Beery VMI) is a measure of visual function. The Beery VMI is a standardized assessment tool designed to evaluate how well individuals can coordinate their visual perception and motor (finger and hand) control. There are three subtests. The main subtest is Visual Motor Integration and the optional subtests are Visual Perception and Motor Coordination. The Beery can be implemented with children 2-18 years. For this study, it will be implemented with children who have the ability to hold a pencil and complete pencil/paper tests.
CVI Range | Aim 2: At enrollment (baseline) and 12 months later
  This study will offer several assessments to test functional vision depending on age and ability level. The CVI Range is a measure of visual function developed by Dr. Christine Roman-Lantzy. The CVI Range is a functional assessment tool used to evaluate the visual abilities of individuals with Cortical/Cerebral Visual Impairment (CVI). The CVI Range helps determine how a person with CVI uses their vision in everyday settings. It is scored on a scale from 1-10 and can be used to assess children from 9 months to 18 years. In this study, it will be used to assess visual function in all participants.
Austin Assessment | Aim 2: At enrollment (baseline) and 12 months later
  The Austin Assessment will be used to measure eye movements and the ability to recognize and match cards with increasing complexity. The test measures search patterns, time to complete, accuracy, and time to initiate the task.
A Developmental NEuroPSYchological Assessment (NEPSY) - Affect Recognition subtest | Aim 2: At enrollment (baseline) and 12 months later
  This study will offer several assessments to test functional vision depending on age and ability level. The NEPSY Affect Recognition subtest measures an aspect of visual function. It designed to assess a child's ability to recognize and interpret facial expressions of emotion. It's part of the Social Perception domain in the NEPSY-II battery. It can be administered to children between 4 to 16 years. It assesses matching faces showing the same emotion, identifying emotions from facial expressions and understanding subtle differences in affect.
Bayley Scale of Infant Development (BSID-IV) | Aim 2: Enrollment (Baseline) and 12 Months later
  The BSID-IV assesses the three neurodevelopmental domains of interest including cognition, language (receptive and expressive) and motor (fine and gross). The BSID will be used to test children 28 months and younger (corrected age if born preterm).
The Peabody Developmental Motor Scales (PDMS) | Aim 2: Enrollment (Baseline) and 12 Months later
  The Peabody Developmental Motor Scales (PDMS-2) is a standardized assessment tool used to evaluate gross and fine motor skills in children from birth through 5 years of age.
Gross Motor Function Measure-66 (GMFM-66) | Aim 2: Enrollment (Baseline) and 12 Months later
  The Gross Motor Function Measure-66 (GMFM-66) is a standardized observational assessment used to evaluate gross motor function in children with cerebral palsy and other motor impairments. It measures changes in gross motor abilities over time or in response to intervention. It can be used for children aged 5 months to 16 years,
The Movement Assessment Battery for Children (MABC) | Aim 2: At enrollment (baseline) and 12 months later
  The Movement Assessment Battery for Children (MABC) is a standardized tool used to assess motor coordination and movement difficulties in children and adolescents aged 3 to 16 years. It is used to identify motor impairments and supports diagnosis of conditions like Developmental Coordination Disorder (DCD).
The Preschool Language Scales- 5th Edition (PLS-5) | Aim 2: Enrollment (Baseline) and 12 Months later
  This study will offer several assessments to test speech and language, depending on age and ability level. The Preschool Language Scales, Fifth Edition (PLS-5) is a standardized assessment tool used to evaluate language development in children from birth through 7 years, 11 months. It assesses both receptive (understanding) and expressive (speaking) language skills.
Rosetti Infant Toddler Language Scale | Aim 2: At enrollment (baseline) and 12 months later
  This study will offer several assessments to test speech and language, depending on age and ability level. The Rossetti Infant-Toddler Language Scale is a criterion-referenced assessment tool used to evaluate communication and language development in children from birth to 3 years of age. It identifies delays in preverbal and verbal communication skills.
Goldman Fristoe Test of Articulation (GFTA) | Aim 2: At enrollment (baseline) and 12 months later
  This study will offer several assessments to test speech and language, depending on age and ability level. For children who present with an articulation deficit, the Goldman Fristoe Test of Articulation will be administered. The GFTA is a standardized assessment used to evaluate articulation skills in individuals aged 2 to 21 years.
The Weschler Preschool & Primary Scale of Intelligence - Fourth Edition (WPPSI-IV) | Aim 2: At enrollment (baseline) and 12 months later
  This study will offer several assessments to test cognition, depending on age and ability level. The Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition (WPPSI-IV) is a standardized cognitive assessment designed for children aged 2 years 6 months to 7 years 7 months. It measures intellectual functioning and helps identify cognitive strengths and weaknesses.
The Leiter International Performance Scale 3 (Leiter 3) | Aim 2: At enrollment (baseline) and 12 months later
  This study will offer several assessments to test cognition, depending on age and ability level. The Leiter International Performance Scale - Third Edition (Leiter-3) is a nonverbal intelligence and cognitive abilities test designed for children aged 3 to 18 years. It assesses nonverbal IQ, attention, memory, and processing speed.

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Harpster, PhD, OTR/L, Principal Investigator — Cincinnati Childrens Hospital Medical Center; Veeral Shah, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided